CLINICAL TRIAL: NCT00563030
Title: Comparison of Granulocyte Subsets in Peripheral Blood After Coronary Bypass Grafting Operations With and Without Use of Cardiopulmonary Bypass
Brief Title: Bands in Peripheral Blood After Coronary Artery Bypass Grafting With and Without Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Maciej M. Kowalik MD, PhD, Medical University of Gdańsk
Other Study IDs: AMG-NKEBN/272/2007
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Granulocyte Immature Forms; Inflammatory Response Syndrome, Systemic
Keywords: Cardiopulmonary bypass; Neutrophils; Coronary artery bypass graft surgery
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood on EDTA vials for automatical morphology analysis and manual blood-smear preparation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients undergoing CABG with CPB
- 2: Patients undergoing off-pump CABG

SUMMARY:
Coronary artery bypass graft (CABG) surgery is associated with reperfusion syndrome and activation of inflammatory reaction (SIRS). These are more exaggerated when cardiopulmonary bypass (CPB) is used.

The aim of the study is to compare signs of SIRS (heart rate, tachypnea or hypocarbia, leukocytosis, hyperpyrexia or hypothermia) and the granulocytes subsets in peripheral blood from patients who underwent CABG surgery with or without use of CPB.

The researchers expect significant differences in SIRS criteria between both groups. If the differences will occur significant, the parameter may be used as candidate variable for a complications prediction model after CABG surgery.

DETAILED DESCRIPTION:
Patients fulfilling inclusion criteria will be asked to sign the consent to participate in the study, the day before operation after routine preoperative anesthesiological evaluation. If included into the study they will be assigned to one of the two study groups - off-pump CABG, or CABG with CPB.

After arrival into the operating theatre 4.5 ml blood will be obtained into EDTA vials from a peripheral venous canula, placed previously for routine anesthesiologic management.

Additional blood samples will be obtained 3, 6, 12, 24 and 48 hours after the operation. Each vial will be immediately labeled with an identification number and submitted into the laboratory, where smear with May-Grunwald-Giemsa staining will be prepared. The smear will be panoptical examined for 400 consecutive leucocytes and assigned to one of the following lines: neutrophils, eosinophils, basophils, monocytes and lymphocytes. Neutrophils will be further divided into: segments, bands, metamyelocytes, myelocytes, promyelocytes, myeloblasts.

The laboratory staff will be blinded for type of operation. Differences in subsets of granulocytes between groups and timepoints wil be analysed as means by appropriate parametric or nonparametric statistical tests.

The SIRS criteria will be refered to:

1. Intraoperative variables: number of distal anastomoses, time of aorta/artery clamping, time of intraoperative hypotension, suction pump use, serum lactates;
2. Postoperative variables: serum CRP, blood products transfusion, chest tube drainage.

ELIGIBILITY:
Inclusion Criteria:

* Elective or urgent CABG with CPB or without (off-pump CABG)
* Signed informed consent

Exclusion Criteria:

* Denied consent
* Signs of infection and/or inflammation (at least 2/4 SIRS criteria)
* Emergency operation
* Organ failure/dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients qualified for elective CABG with or without cardiopulmonary bypass. If possible, patient will be matched by age, sex, left ventricle ejection fraction, number of grafts, and major comorbidities (diabetes mellitus, arteriosclerosis).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
percentage of immature forms of neutrophils in peripheral blood | first 48 hours after operation

SECONDARY OUTCOMES:
clinical signs of SIRS: heart rate, temperature, pCO2, respiratory rate (as applicable), total white blood cells | first 48 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: Maciej M Kowalik, MD, PhD, Study Director — Medical University of Gdańsk, Dept. of Cardiac Anesthesiology
Locations (1):
- Medical University of Gdańsk, Dept. of Cardiac Anesthesiology, Gdansk, Poland

REFERENCES:
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Santa Ursula Tolosa JA, Criado A, Garcia del Valle S, Pensado A, Barbolla L, Carmona Aurioles JA. [Changes in total and differential leukocyte counts during heart surgery with extracorporeal circulation]. Rev Esp Anestesiol Reanim. 1991 Mar-Apr;38(2):94-7. Spanish. PMID 1876745
- [Background] Orr Y, Taylor JM, Bannon PG, Geczy C, Kritharides L. Circulating CD10-/CD16low neutrophils provide a quantitative index of active bone marrow neutrophil release. Br J Haematol. 2005 Nov;131(4):508-19. doi: 10.1111/j.1365-2141.2005.05794.x. PMID 16281943
- [Background] Orr Y, Wilson DP, Taylor JM, Bannon PG, Geczy C, Davenport MP, Kritharides L. A kinetic model of bone marrow neutrophil production that characterizes late phenotypic maturation. Am J Physiol Regul Integr Comp Physiol. 2007 Apr;292(4):R1707-16. doi: 10.1152/ajpregu.00627.2006. Epub 2006 Dec 21. PMID 17185405
- See also: home page of Dept. of Cardiac Anesthesiology, Medical University of Gdańsk — http://www.amg.gda.pl/uczelnia/informator/jednostka.php?id=327